CLINICAL TRIAL: NCT04121455
Title: Single-arm, Dose-escalation Phase 1/2 Study of Olaptesed Pegol (NOX-A12) in Combination With Irradiation in Inoperable or Partially Resected First-line Glioblastoma Patients With Unmethylated MGMT Promoter With a Multiple-arm Expansion Group
Brief Title: Glioblastoma Treatment With Irradiation and Olaptesed Pegol (NOX-A12) in MGMT Unmethylated Patients
Acronym: GLORIA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNOXA12C401; 2024-510964-21-00 (EU CTIS Number); 2018-004064-62 (EudraCT Number)
Record Dates: First submitted 2019-09-25; First posted 2019-10-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; NOX-A12; Olaptesed pegol; Spiegelmer; Stromal cell-derived factor-1 (SDF-1); CXCL12; Radiation; MGMT promoter; Brain tumor; Radiotherapy; Brain cancer; Tumor microenvironment; Bevacizumab
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — NOX-A12; Radiotherapy; Bevacizumab; pembrolizumab; Temozolomide

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation (sequential) followed by a multiple-arm expansion group (parallel)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1: 200 mg Olaptesed pegol + Radiotherapy (Experimental): olaptesed pegol weekly for 26 weeks administered i.v. by continuous infusion plus radiotherapy during weeks 1-6
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy
- Cohort 2: 400 mg Olaptesed pegol + Radiotherapy (Experimental): olaptesed pegol weekly for 26 weeks administered i.v. by continuous infusion plus radiotherapy during weeks 1-6
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy
- Cohort 3: 600 mg Olaptesed pegol + Radiotherapy (Experimental): olaptesed pegol weekly for 26 weeks administered i.v. by continuous infusion plus radiotherapy during weeks 1-6
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy
- Expansion group, Arm A: 600 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab (Experimental): olaptesed pegol weekly for 26 weeks administered i.v. by continuous infusion, bevacizumab every two weeks for 26 weeks plus radiotherapy during weeks 1-6, incompletely or not resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy; Drug: Bevacizumab
- Expansion group, Arm B: 600 mg Olaptesed pegol + Radiotherapy (Experimental): olaptesed pegol weekly for 26 weeks administered i.v. by continuous infusion plus radiotherapy during weeks 1-6, completely resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy
- Expansion group, Arm C: 600 mg Olaptesed pegol + Radiotherapy + 200 mg Pembrolizumab (Experimental): olaptesed pegol weekly for 26 weeks administered i.v. by continuous infusion, pembrolizumab every three weeks for 26 weeks plus radiotherapy during weeks 1-6, incompletely resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy; Drug: Pembrolizumab
- Expansion group, Arm D: 200 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab (Experimental): olaptesed pegol i.v. by continuous infusion, bevacizumab every two weeks plus radiotherapy during weeks 1-6, until progression or intolerable toxicity (patients with disease progression may continue treatment with all assessments if deemed appropriate by the investigator), incompletely resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy; Drug: Bevacizumab
- Expansion group, Arm E: 400 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab (Experimental): olaptesed pegol i.v. by continuous infusion, bevacizumab every two weeks plus radiotherapy during weeks 1-6, until progression or intolerable toxicity (patients with disease progression may continue treatment with all assessments if deemed appropriate by the investigator), incompletely resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy; Drug: Bevacizumab
- Expansion group, Arm F: 600 mg Olaptesed pegol + Radiotherapy + 10 mg/kgBevacizumab (Experimental): olaptesed pegol i.v. by continuous infusion, bevacizumab every two weeks plus radiotherapy during weeks 1-6, until progression or intolerable toxicity (patients with disease progression may continue treatment with all assessments if deemed appropriate by the investigator), incompletely resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy; Drug: Bevacizumab
- Expansion group, Arm G: 600 mg Olaptesed pegol + Radiotherapy (Experimental): olaptesed pegol i.v. by continuous infusion, bevacizumab every two weeks plus radiotherapy during weeks 1-6, until progression or intolerable toxicity (patients with disease progression may continue treatment with all assessments if deemed appropriate by the investigator), incompletely resected patients
  Interventions: Drug: Olaptesed pegol; Radiation: Radiotherapy
- Expansion group, Arm H: Standard of care - Temozolomide + Radiotherapy (Active Comparator): oral treatment up to 35 weeks according to current SPC
  Interventions: Radiation: Radiotherapy; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Olaptesed pegol — Olaptesed pegol continuous i.v. administration
  Other Names: NOX-A12
  Arms: Cohort 1: 200 mg Olaptesed pegol + Radiotherapy; Cohort 2: 400 mg Olaptesed pegol + Radiotherapy; Cohort 3: 600 mg Olaptesed pegol + Radiotherapy; Expansion group, Arm A: 600 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab; Expansion group, Arm B: 600 mg Olaptesed pegol + Radiotherapy; Expansion group, Arm C: 600 mg Olaptesed pegol + Radiotherapy + 200 mg Pembrolizumab; Expansion group, Arm D: 200 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab; Expansion group, Arm E: 400 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab; Expansion group, Arm F: 600 mg Olaptesed pegol + Radiotherapy + 10 mg/kgBevacizumab; Expansion group, Arm G: 600 mg Olaptesed pegol + Radiotherapy
Radiation: Radiotherapy — Radiotherapy in weeks 1-6; cumulative dose of 60 Gy in 2 Gy fractions
Drug: Bevacizumab — Bevacizumab every 2 weeks i.v. infusion
  Arms: Expansion group, Arm A: 600 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab; Expansion group, Arm D: 200 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab; Expansion group, Arm E: 400 mg Olaptesed pegol + Radiotherapy + 10 mg/kg Bevacizumab; Expansion group, Arm F: 600 mg Olaptesed pegol + Radiotherapy + 10 mg/kgBevacizumab
Drug: Pembrolizumab — Pembrolizumab every 3 weeks i.v. for 26 weeks
  Other Names: KEYTRUDA
  Arms: Expansion group, Arm C: 600 mg Olaptesed pegol + Radiotherapy + 200 mg Pembrolizumab
Drug: Temozolomide (TMZ) — oral treatment according to current SPC
  Arms: Expansion group, Arm H: Standard of care - Temozolomide + Radiotherapy

SUMMARY:
The purpose of this study is to obtain first, exploratory information on the safety and efficacy of (i) olaptesed pegol in combination with radiation therapy in patients with newly diagnosed glioblastoma of unmethylated MGMT promoter status either not amenable to resection (biopsy only) or after incomplete tumor resection, and (ii) olaptesed pegol in combination with radiation therapy and bevacizumab in patients with newly diagnosed glioblastoma of unmethylated MGMT promoter status either not amenable to resection (biopsy only) or after incomplete or complete tumor resection.

Further arms are included (i) to establish safety for the combination of olaptesed pegol at three different doses in addition to radiotherapy and bevacizumab, (ii) to explore the benefit of combining olaptesed pegol at different dose levels with bevacizumab in order to define the doses to move forward into a subsequent randomized dose-finding study, (iii) to explore the contribution of the therapy components olaptesed pegol and bevacizumab to patient benefit and (iv) to put the clinical outcome of these treatment regimens into perspective with the standard of care treatment with temozolomide and radiotherapy.

ELIGIBILITY:
Inclusion Criteria Dose Escalation Cohorts:

1. Written informed consent
2. Age ≥18 years
3. Patient agreement to diagnostic and scientific work-up of glioblastoma tissue obtained during the preceding surgery or biopsy
4. Patient agrees to subcutaneous port implantation
5. Newly diagnosed, histologically confirmed, supratentorial WHO grade IV glioblastoma
6. Status post biopsy or incomplete resection
7. Unmethylated MGMT promoter status
8. Maximum Eastern Cooperative Oncology Group (ECOG) score 2
9. Estimated minimum life expectancy 3 months
10. Stable or decreasing dose of corticosteroids during the week prior to inclusion
11. The following laboratory parameters should be within the ranges specified:

    * Total bilirubin ≤ 1.5 x upper limit normal (ULN)
    * Creatinine ≤ 1.5 x ULN or glomerular filtration rate ≥ 60 mL/min/1.73m²
    * ALT (alanine transaminase) ≤ 3 x ULN
    * AST (aspartate transaminase) ≤ 3 x ULN
12. Female patients of child-bearing potential must have a negative serum pregnancy test within 21 days prior to enrollment and agree to use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly such as contraceptive implants, vaginal rings, sterilization, or sexual abstinence)" during and for 3 months following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations)
13. Male patients must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a FCBP

Inclusion Criteria Expansion Group Arms A, B and C:

1. Written informed consent
2. Age ≥ 18 years
3. Patient agreement to diagnostic and scientific work-up of glioblastoma tissue obtained during the preceding surgery or biopsy (e.g., MGMT promoter analysis, cytogenetic markers such as IDH-1 mutations, etc.)
4. Patient agrees to subcutaneous port implantation
5. Newly diagnosed, histologically confirmed, supratentorial WHO grade IV glioblastoma
6. a) Status post biopsy or incomplete (detectable residual tumor as per postoperative T1-weighted, contrast-enhanced MRI scan) or complete resection (Arm A) OR b) Status post complete resection (Arm B) OR c) Status post complete or incomplete resection (circumscribed enhancing tumor ≤ 5.0 cm in largest diameter as per postoperative T1-weighted, contrast-enhanced MRI scan) (Arm C)
7. Unmethylated MGMT promoter status
8. Maximum Eastern Cooperative Oncology Group (ECOG) score 2
9. Estimated minimum life expectancy 3 months
10. Stable or decreasing dose of corticosteroids during the week prior to inclusion
11. The following laboratory parameters should be within the ranges specified:

    * Total bilirubin ≤ 1.5 x upper limit normal (ULN)
    * Creatinine ≤ 1.5 x ULN or glomerular filtration rate ≥ 60 mL/min/1.73m²
    * ALT (alanine transaminase) ≤ 3 x ULN
    * AST (aspartate transaminase) ≤ 3 x ULN
12. Female patients of child-bearing potential must have a negative serum pregnancy test within 21 days prior to enrollment and agree to use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly such as contraceptive implants, vaginal rings, sterilization, or sexual abstinence) during and for 3 months (6 months Arm A, 4 months Arm C) following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations)
13. Male patients must use an effective barrier method of contraception during study and for 3 months (6 months Arm A, 4 months Arm C) following the last dose if sexually active with a FCBP

Inclusion Criteria Expansion Group Arms D, E, F, G, and H:

1. Written informed consent
2. Age ≥ 18 years
3. Patient agreement to diagnostic and scientific work-up of glioblastoma tissue obtained during the preceding surgery (e.g., MGMT promoter analysis, cytogenetic markers such as IDH-1 mutations, etc.)
4. Patient agrees to subcutaneous port implantation
5. Newly diagnosed, histologically confirmed, supratentorial WHO grade 4 glioblastoma, IDH-wildtype according to the 2021 World Health Organization Criteria for CNS tumors
6. Status post incomplete resection (detectable residual tumor as per postoperative T1-weighted, contrast-enhanced MRI scan)
7. Unmethylated MGMT promoter status
8. Maximum Eastern Cooperative Oncology Group (ECOG) score 2
9. Estimated minimum life expectancy 3 months
10. Stable or decreasing dose of corticosteroids during the week prior to inclusion
11. The following laboratory parameters should be within the ranges specified:

    * Total bilirubin ≤ 1.5 x upper limit normal (ULN)
    * Body surface area (BSA) adjusted glomerular filtration rate (GFR) ≥ 60 mL/min (BSA-adjusted eGFR CKD-EPI (mL/min) = [eGFR CKD-EPI (mL/min/1.73 m²) x BSA (m²)]/ 1.73; BSA calculated by Du Bois formula)
    * Alanine transaminase (ALT) ≤ 3 x ULN
    * Aspartate transaminase (AST) ≤ 3 x ULN
    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L and platelet count ≥ 100 x 10^9/L
12. Female patients of child-bearing potential (FCBP) must have a negative serum pregnancy test within 21 days prior to enrollment and agree to use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly such as contraceptive implants, vaginal rings, sterilization, or sexual abstinence) during and for 6 months following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations)
13. Male patients must use an effective barrier method of contraception during study and for 6 months following the last dose if sexually active with a FCBP

Exclusion Criteria Dose Escalation Cohorts:

1. Inability to understand and collaborate throughout the study or inability or unwillingness to comply with study requirements
2. Participation in any clinical research study with administration of an investigational drug or therapy within 30 days from screening visit or observation period of competing studies
3. Contra-indication or known hypersensitivity to MRI contrast agents, olaptesed pegol or polyethylene glycol
4. Cytostatic therapy (chemotherapy) within the past 5 years
5. History of other cancers (except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient was disease-free for ≥ 5 years)
6. Clinically significant or uncontrolled cardiovascular disease
7. Prior radiotherapy to the head
8. Any other previous or concomitant experimental glioblastoma treatments
9. Placement of Gliadel® wafer, seeds, or ferromagnetic nanoparticles
10. Pregnancy or lactation
11. Uncontrolled intercurrent illness; patients must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations
12. Treatment not initiated within 6 weeks after first biopsy or surgery of glioblastoma
13. Prior enrolment into this study

Exclusion Criteria Expansion Group Arms A and B:

1. Inability to understand and collaborate throughout the study or inability or unwillingness to comply with study requirements
2. Participation in any clinical research study with administration of an investigational drug or therapy within 30 days from screening visit or observation period of competing studies
3. Contra-indication or known hypersensitivity to MRI contrast agents, bevacizumab (Arm A only) olaptesed pegol or polyethylene glycol
4. Planned hypofractionated radiotherapy
5. Cytostatic therapy (chemotherapy) within the past 5 years
6. History of other cancers (except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient was disease-free for ≥ 5 years)
7. Secondary malignancy which is currently active
8. Clinically significant or uncontrolled cardiovascular disease, including

   * Myocardial infarction in the previous 12 months
   * Uncontrolled angina
   * Congestive heart failure (New York Heart Association functional classification of ≥2)
   * Diagnosed or suspected congenital long QT syndrome
   * QTc prolongation on an electrocardiogram prior to entry (QTc(Bazett) >470 ms)
   * Uncontrolled hypertension (blood pressure ≥ 160/95 mmHg)
   * Heart rate <50/min on the baseline electrocardiogram
   * History of ventricular arrhythmias of any clinically significant type (such as ventricular tachycardia, ventricular fibrillation or torsades de pointes)
   * Cerebrovascular accident
9. Prior radiotherapy to the head
10. Any other previous or concomitant experimental glioblastoma treatments
11. Placement of Gliadel® wafer, seeds, or ferromagnetic nanoparticles
12. Patients with a history of arterial or venous thrombosis (or any other disease) requiring permanent intake of anticoagulants (Arm A only)
13. Pregnancy or lactation
14. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), diabetes mellitus, or subjects with either of the following: fasting blood glucose (FBG defined as fasting for at least 8 hours) ≥ 200 mg/dL (7.0 mmol/L), or HbA1c ≥ 8%, chronic renal disease, pancreatitis, chronic pulmonary disease, auto-immune diseases, or psychiatric illness/social situations that would limit compliance with study requirements. Patients must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations
15. Prolongation of coagulation factors ≥ 2.5 x ULN (Arm A only)
16. Treatment not initiated within 6 weeks after first biopsy or surgery of glioblastoma
17. Prior enrolment into this study

Exclusion Criteria Expansion Group Arms C:

1. Inability to understand and collaborate throughout the study or inability or unwillingness to comply with study requirements
2. Participation in any clinical research study with administration of an investigational drug or therapy within 30 days from screening visit or observation period of competing studies
3. Contra-indication or known hypersensitivity to MRI contrast agents olaptesed pegol or polyethylene glycol or pembrolizumab (≥ Grade 3)
4. Biopsy-only of GBM with less than 20% of tumor removed
5. Presence of extracranial metastatic or leptomeningeal disease
6. Severe hypersensitivity (≥ Grade 3) to other monoclonal antibodies
7. Receiving immunosuppressive therapy
8. Previous or current treatment with an anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PDL2 agent
9. Planned hypofractionated radiotherapy
10. Cytostatic therapy (chemotherapy) within the past 5 years
11. History of other cancers or secondary malignancy which is currently active (except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient was disease-free for ≥ 5 years)
12. Clinically significant or uncontrolled cardiovascular disease, including

    * Myocardial infarction in the previous 12 months
    * Uncontrolled angina
    * Congestive heart failure (New York Heart Association functional classification of ≥2)
    * Diagnosed or suspected congenital long QT syndrome
    * QTc prolongation on an electrocardiogram prior to entry (QTc(Bazett) >470 ms)
    * Uncontrolled hypertension (blood pressure ≥ 160/95 mmHg)
    * Heart rate <50/min on the baseline electrocardiogram
    * History of ventricular arrhythmias of any clinically significant type (such as ventricular tachycardia, ventricular fibrillation or torsades de pointes)
    * Cerebrovascular accident
13. Prior radiotherapy to the head
14. Evidence of acute intracranial / intra-tumoral hemorrhage
15. Any other previous or concomitant experimental glioblastoma treatments
16. Placement of Gliadel® wafer, seeds, or ferromagnetic nanoparticles
17. Pregnancy or lactation
18. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), diabetes mellitus, or subjects with either of the following: fasting blood glucose (FBG defined as fasting for at least 8 hours) ≥ 200 mg/dL (7.0 mmol/L), or HbA1c ≥ 8%, chronic renal disease, pancreatitis, chronic pulmonary disease, auto-immune diseases or psychiatric illness/social situations that would limit compliance with study requirements. Patients must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations.
19. Received a live vaccine within 30 days prior to the first dose of study drug.
20. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Previously treated brain metastases may participate provided these remain stable
21. Known history of HIV infection, hepatitis B or hepatitis C infection
22. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
23. History of (non-infectious) pneumonitis / interstitial lung disease that required steroids or current pneumonitis / interstitial lung disease
24. Immunodeficiency diagnosis or receiving chronic systemic steroid therapy (exceeding 10 mg daily of prednisone) or any other form of immunosuppressive therapy
25. High dose of corticosteroids (≥ 4mg/day of dexamethasone or equivalent for at least 3 consecutive days) within two weeks prior to the first dose of study drug
26. Treatment not initiated within 6 weeks after first biopsy or surgery of glioblastoma
27. Prior enrolment into this study

Exclusion Criteria Expansion Group Arms D, E, F, G and H:

1. Patients with tumors harboring IDH mutations
2. Inability to understand and collaborate throughout the study or inability or unwillingness to comply with study requirements
3. Participation in any clinical research study with administration of an investigational drug or therapy within 30 days prior to screening visit or observation period of competing studies
4. Contra-indication or known hypersensitivity to MRI contrast agents, bevacizumab, olaptesed pegol or polyethylene glycol
5. Planned hypofractionated radiotherapy
6. Chemotherapy (cytotoxic/cytostatic) within the past 5 years
7. History of other cancers (except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient was disease-free for ≥ 5 years)
8. Secondary malignancy which is currently active
9. Clinically significant or uncontrolled cardiovascular disease, including

   * Myocardial infarction in the previous 12 months
   * Uncontrolled angina
   * Congestive heart failure (New York Heart Association functional classification of ≥2)
   * Diagnosed or suspected congenital long QT syndrome
   * QTc prolongation on the electrocardiogram prior to inclusion (QTc(Bazett) >470 ms)
   * Uncontrolled hypertension (blood pressure ≥ 160/95 mmHg)
   * Heart rate <50/min on the electrocardiogram prior to inclusion
   * History of ventricular arrhythmias of any clinically significant type (such as ventricular tachycardia, ventricular fibrillation or torsades de pointes)
   * Cerebrovascular accident
10. Prior radiotherapy to the head
11. Any other previous or concomitant experimental glioblastoma treatments
12. Placement of Gliadel® wafer, seeds, or ferromagnetic nanoparticles
13. Patients with a history of arterial or venous thrombosis (or any other disease) requiring permanent intake of anticoagulants
14. Pregnancy or lactation
15. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), diabetes mellitus, or patients with either of the following: fasting blood glucose (FBG defined as fasting for at least 8 hours) ≥ 200 mg/dL (7.0 mmol/L), or HbA1c ≥ 8%, chronic renal disease, pancreatitis, chronic pulmonary disease, auto-immune diseases or psychiatric illness/social situations that would limit compliance with study requirements. Patients must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations.
16. Prolongation of coagulation factors ≥ 2.5 x ULN
17. Treatment not initiated within 6 weeks after surgery of glioblastoma
18. Prior enrolment into this study
19. History of hypersensitivity to dacarbazine (DTIC)
20. History of hypersensitivity reaction (such as urticaria, allergic reaction including anaphylaxis, toxic epidermal necrolysis, and Stevens-Johnson syndrome) to temozolomide or any of its components
21. Severe myelosuppression (ANC <1.5 x 10^9/L and platelet count <100 x 10^9/L)
22. Major surgery within 28 days prior to treatment start
23. Non-healing wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety - Number of patients with treatment-related adverse events as assessed by CTCAE | through study completion, an average of 3 years
  Number of patients with treatment-related adverse events as assessed by CTCAE

SECONDARY OUTCOMES:
Efficacy - progression free survival at 6 months (PFS-6) | 6 months
  Progression free survival at 6 months (PFS-6) in %
Efficacy - Median progression-free survival (mPFS) | until end of treatment, an average 1 year
  Median progression-free survival (mPFS) in months
Efficacy - Median overall survival (mOS) | through study completion, an average of 3 years
  Median overall survival (mOS) in months
Efficacy - Landmark overall survival at 18 months (OS18) | 18 months
Overall response rate (ORR) | through study completion, an average of 3 years
Plasma level of olaptesed pegol | 9 weeks after treatment start
  concentration of olaptesed pegol in plasma in µmol/L
Quality of Life (QoL) EORTC QLQ-C30 Module | through study completion, an average of 3 years
  Quality of Life measures are recorded according to EORTC QLQ30 module, which is validated for cancer patients in general and measured as a unit of scale. This is a standard tool for assessing patient reported quality of Life along time during treatment.
Quality of Life (QoL) EORTC QLQ BN-20 Module | through study completion, an average of 3 years
  Quality of Life measures are recorded according to EORTC QLQ BN-20 module, which is validated for brain tumor patients and measured as a unit of scale. This is a standard tool for assessing patient reported quality of Life along time during treatment.
Efficacy - Tumor vascularization as per vascular MRI | through study completion, an average of 3 years
  Changes from baseline in tumor vascularization over time as %cerebral blood volume
Neurologic functions as measured by the NANO scale | 24 months
  Change from baseline in neurologic performance scores by Neurologic Assessment in Neuro-Oncology (NANO) scale as an objective and quantifiable metric of neurologic function evaluable during a routine office examination. The NANO Scale evaluates 9 major domains of neurologic function, with each domain being scored on a range from 0 to 2 or 3.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Klinik und Poliklinik für Neurologie Schwerpunkt Klinische Neuroonkologie, Bonn
  - Klinik für Neurologie, Essen
  - Klinik für Strahlentherapie und Radioonkologie, Leipzig
  - Klinik für Strahlentherapie und Radioonkologie, Mannheim
  - Klinik für Neurologie mit Institut für Translationale Neurologie, Münster
  - Abteilung Neurologie mit interdisziplinärem Schwerpunkt Neuroonkologie, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided